CLINICAL TRIAL: NCT05029232
Title: Comprehensive Study of Duchenne Muscular Dystrophy at Sohag University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nehal Samy Abdo, Assistant lecturer of pediatric. sohag university hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-21-07-21
Record Dates: First submitted 2021-07-14; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Thyroid Function Tests; Electromyography; Neural Conduction; Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ambulant patient with DMD (Active Comparator): patient that walk alone or with minor assist
  Interventions: Diagnostic Test: MLPA for duchenne
- non ambulant patient with DMD (Active Comparator): patient need wheel chair
  Interventions: Diagnostic Test: MLPA for duchenne

INTERVENTIONS:
Diagnostic Test: MLPA for duchenne — MLPA test for genetic testing to detect gene affection in DMD , and other tests for confirmation and follow up
  Other Names: muscle enzymes; thyroid function; EMG , nerve conduction for limbs; echocardiography , MRI brain , IQ test

SUMMARY:
Muscular dystrophies are a heterogenous group of inherited muscular disorders characterized by progressive muscle weakness. Historically, these disorders are difficult to treat. In the last three decades, there is a great progress in molecular and genetic basis of these disorders; early diagnosis is achievable with proper clinical recognition and advanced genetic testing .Duchenne Muscular Dystrophy (DMD) is a neuromuscular muscular X-linked recessive disorders that belong to a group of disorders known as dystrophinopathies. DMD characterized by a progressive degeneration of skeletal muscles, with symptoms that manifest early, at around 3 years, causing loss of ambulation within the 13 years of life, followed by cardiac complication (e.g., dilated cardiomyopathy and arrhythmia) and respiratory disorders, including chronic respiratory failure. The unique medical treatment available is steroid therapy, which appears to prolong walking capacity by at least two years. Thus, besides medical treatment, the physical therapy in multidisciplinary care is imperative for alleviating muscle atrophy, skeletal deformities, and motor function deterioration.

ELIGIBILITY:
Inclusion Criteria:

1. age of onset between 3- and 18-year-old
2. typical clinical manifestation of Duchenne muscular dystrophy
3. clinical manifestation confirmed by specific biochemical analysis or by genetic testing who presented to pediatric department and neurology outpatient clinic during the period of study.

Exclusion Criteria:

1. children with another congenital muscular dystrophy
2. children with other types of myopathies
3. presence of CNS disorders such as brain insult & spinal muscular atrophy
4. female gender

Ages: 3 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
change in dystrophine gene mutation | within six months
  MLPA test
change in MRI findings in DMX patient from normal | within six months
  by MRI brain
change in cardiac function in DMD patient | within six months
  by Echocardiography to detect EF, FS
change in thyroid function in DMD patient | within six months
  by thyroid function test
change in cognitive function in DMD patients | within six months
  by Stanford IQ test

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Birnkrant DJ, Bushby K, Bann CM, Apkon SD, Blackwell A, Brumbaugh D, Case LE, Clemens PR, Hadjiyannakis S, Pandya S, Street N, Tomezsko J, Wagner KR, Ward LM, Weber DR; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 1: diagnosis, and neuromuscular, rehabilitation, endocrine, and gastrointestinal and nutritional management. Lancet Neurol. 2018 Mar;17(3):251-267. doi: 10.1016/S1474-4422(18)30024-3. Epub 2018 Feb 3. PMID 29395989
- [Background] Birnkrant DJ, Bushby K, Bann CM, Alman BA, Apkon SD, Blackwell A, Case LE, Cripe L, Hadjiyannakis S, Olson AK, Sheehan DW, Bolen J, Weber DR, Ward LM; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 2: respiratory, cardiac, bone health, and orthopaedic management. Lancet Neurol. 2018 Apr;17(4):347-361. doi: 10.1016/S1474-4422(18)30025-5. Epub 2018 Feb 3. PMID 29395990
- [Background] Giliberto F, Radic CP, Luce L, Ferreiro V, de Brasi C, Szijan I. Symptomatic female carriers of Duchenne muscular dystrophy (DMD): genetic and clinical characterization. J Neurol Sci. 2014 Jan 15;336(1-2):36-41. doi: 10.1016/j.jns.2013.09.036. Epub 2013 Oct 5. PMID 24135430